CLINICAL TRIAL: NCT01419717
Title: Open-Label Access Protocol of Denosumab for Subjects With Advanced Cancer
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Amgen (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 20110113
Record Dates: First submitted 2011-08-04; First posted 2011-08-18 (Estimated); Results first posted 2019-09-09 (Actual); Last update posted 2019-09-24 (Actual); Status verified 2019-09

CONDITIONS: Bone Metastases in Men With Hormone-Refractory Prostate Cancer; Bone Metastases in Subjects With Advanced Breast Cancer
Keywords: cancer; bone metastases; breast cancer; prostate cancer
MeSH Terms: conditions — Neoplasms; Breast Neoplasms; Prostatic Neoplasms | interventions — Denosumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Denosumab (Experimental): Participants received 120 milligrams of denosumab injected subcutaneously every 4 weeks until denosumab was approved and available for sale.
  Interventions: Drug: Denosumab

INTERVENTIONS:
Drug: Denosumab — Administered by subcutaneous injection every 4 weeks (Q4W)
  Other Names: Xgeva

SUMMARY:
This trial will facilitate access to denosumab for adults with advanced cancer who have participated in a denosumab phase 3 study until denosumab is approved and available for sale.

ELIGIBILITY:
Inclusion Criteria:

* Subject was previously enrolled in a denosumab phase 3 study and participated in the Open-label Extension portion of that study.
* Subject or subject's legally acceptable representative has provided informed consent.

Exclusion Criteria:

* Subject is of child bearing potential and planning to become pregnant within 7 months after the end of treatment.
* Subject is of child bearing potential and is not willing to use, in combination with her partner, two highly effective methods of contraception during treatment and for 7 months after the end of treatment.
* Subject has known sensitivity to any of the products to be administered during dosing.
* Subject will not be available for protocol required study visits or procedures, to the best of the subject and investigator's knowledge.
* Subject has any kind of disorder that, in the opinion of the investigator, may compromise the ability of the subject to give written informed consent and/or to comply with all required study procedures.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 129 (Actual)
Dates: Start 2011-11-22 (Actual); Primary Completion 2018-08-10 (Actual); Study Completion 2018-08-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: MD, Study Director — Amgen
Locations (55):
- Argentina (4):
  - Research Site, Capital Federal, Buenos Aires
  - Research Site, Quilmes, Buenos Aires
  - Research Site, Córdoba, Córdoba Province
  - Research Site, Rosario, Santa Fe Province
- Research Site, Vienna, Austria
- Research Site, Namur, Belgium
- Brazil (6):
  - Research Site, Porto Alegre, Rio Grande do Sul
  - Research Site, Santo André, São Paulo
  - Research Site, São Paulo, São Paulo
  - Research Site, Sorocaba, São Paulo
  - Research Site, Rio de Janeiro
  - Research Site, São Paulo
- Czechia (3):
  - Research Site, Kroměříž
  - Research Site, Olomouc
  - Research Site, Prague
- Research Site, Saint-Cloud, France
- Hungary (2):
  - Research Site, Debrecen
  - Research Site, Dombóvár
- Israel (4):
  - Research Site, Haifa
  - Research Site, Rehovot
  - Research Site, Tel Aviv
  - Research Site, Ẕerifin
- Italy (2):
  - Research Site, Meldola (FC)
  - Research Site, Sora
- Japan (7):
  - Research Site, Kure-shi, Hiroshima
  - Research Site, Kagoshima, Kagoshima-ken
  - Research Site, Isehara-shi, Kanagawa
  - Research Site, Osaka, Osaka
  - Research Site, Kitaadachi-gun, Saitama
  - Research Site, Chuo-ku, Tokyo
  - Research Site, Tokyo
- Latvia (2):
  - Research Site, Daugavpils
  - Research Site, Riga
- Lithuania (2):
  - Research Site, Kaunas
  - Research Site, Vilnius
- Research Site, Panama City, Panama
- Research Site, Lima, Peru
- Poland (6):
  - Research Site, Bialystok
  - Research Site, Bydgoszcz
  - Research Site, Gdansk
  - Research Site, Lublin
  - Research Site, Poznan
  - Research Site, Warsaw
- Russia (7):
  - Research Site, Arkhangelsk
  - Research Site, Chelyabinsk
  - Research Site, Krasnogorsky District
  - Research Site, Moscow
  - Research Site, Obninsk
  - Research Site, Omsk
  - Research Site, Saint Petersburg
- Research Site, Pretoria, South Africa
- Spain (3):
  - Research Site, Seville, Andalusia
  - Research Site, Valencia, Valencia
  - Research Site, Madrid
- Research Site, Lviv, Ukraine

IPD SHARING:
Plan to Share IPD: Yes
De-identified individual patient data for variables necessary to address the specific research question in an approved data sharing request
Supporting Information: Study Protocol, SAP, ICF, CSR
Time Frame: Data sharing requests relating to this study will be considered beginning 18 months after the study has ended and either 1) the product and indication have been granted marketing authorization in both the US and Europe or 2) clinical development for the product and/or indication discontinues and the data will not be submitted to regulatory authorities. There is no end date for eligibility to submit a data sharing request for this study.
Access Criteria: Qualified researchers may submit a request containing the research objectives, the Amgen product(s) and Amgen study/studies in scope, endpoints/outcomes of interest, statistical analysis plan, data requirements, publication plan, and qualifications of the researcher(s). In general, Amgen does not grant external requests for individual patient data for the purpose of re-evaluating safety and efficacy issues already addressed in the product labelling. Requests are reviewed by a committee of internal advisors. If not approved, a Data Sharing Independent Review Panel will arbitrate and make the final decision. Upon approval, information necessary to address the research question will be provided under the terms of a data sharing agreement. This may include anonymized individual patient data and/or available supporting documents, containing fragments of analysis code where provided in analysis specifications. Further details are available at the link below.
URL: https://www.amgen.com/datasharing

REFERENCES:
- See also: AmgenTrials clinical trials website — http://www.amgentrials.com

RESULTS

PARTICIPANT FLOW:
Recruitment Details: This study was conducted at 65 centers in Europe, Latin America, Japan, and South Africa. Participants were enrolled from 22 November 2011 to 27 October 2014.
Groups:
- Denosumab: Participants were offered 120 milligrams of denosumab injected subcutaneously every 4 weeks until denosumab was approved and available for sale.
Period: Overall Study
Arm/Group | Denosumab
Started | 129
Received Denosumab | 128
Completed | 4
Not Completed | 125
Not completed — Protocol-specified Criteria | 62
Not completed — Adverse Event | 19
Not completed — Death | 17
Not completed — Withdrawal by Subject | 10
Not completed — Disease Progression | 9
Not completed — Other | 4
Not completed — Lost to Follow-up | 2
Not completed — Administrative Decision | 1
Not completed — Noncompliance | 1

BASELINE CHARACTERISTICS:
Arm/Group | Denosumab
Number analyzed (Participants) | 129
Age, Continuous [Mean (Standard Deviation); unit: years] | 65.74 (11.48)
Age, Customized [Count of Participants; unit: Participants]
  18 - 64 years | 60
  65 - 74 years | 36
  75 - 84 years | 28
  ≥ 85 years | 5
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 97
  Male | 32
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 28
  Not Hispanic or Latino | 101
  Unknown or Not Reported | 0
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  White | 103
  Asian | 15
  Black or African American | 6
  Other | 4
  Unknown | 1

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Adverse Events
Description: An adverse event (AE) is defined as any untoward medical occurrence in a clinical trial participant. The event does not necessarily have a causal relationship with study treatment.
  Each AE was graded for severity according to the Common Terminology Criteria for Adverse Events (CTCAE) version 3.0, where Grade 1 = Mild AE Grade 2 = Moderate AE Grade 3 = Severe AE Grade 4 = Life-threatening or disabling AE Grade 5 = Death related to AE. Treatment-related adverse events (TRAEs) includes events for which the investigator indicated there was a reasonable possibility they may have been caused by investigational product.
Time Frame: From first dose of denosumab in Study 20110113 to end of study; median (minimum, maximum) time on study was 13.93 (0.0, 74.7) months.
Population: All participants who received at least one dose of denosumab in study 20110113
Measure: Count of Participants; unit: Participants
Arm/Group | Denosumab
Number analyzed (Participants) | 128
Participants
  All adverse events | 98
  Serious adverse events | 45
  AE leading to discontinuation of denosumab | 28
  AE leading to discontinuation from study | 22
  Fatal adverse events | 18
  AE grade 3, 4, or 5 | 46
  Treatment-related adverse event | 26
  Treatment-related serious adverse event | 10
  TRAE leading to discontinuation of denosumab | 18
  TRAE leading to discontinuation from study | 16
  Treatment-related fatal adverse events | 0
  Treatment-related AE grade 3, 4, or 5 | 8

2. Secondary Outcome: Number of Participants With Anti-denosumab Binding Antibodies
Description: A blood sample was collected at the end of study visit for the measurement of anti-denosumab binding antibodies.
Time Frame: Assessed at end of study; the median (minimum, maximum) time on study for all enrolled participants was 13.9 (0.0, 74.7) months.
Population: Participants who received at least 1 dose of denosumab in study 20110113 and with at least 1 antibody sample tested.
Measure: Count of Participants; unit: Participants
Arm/Group | Denosumab
Number analyzed (Participants) | 86
Participants | 0

ADVERSE EVENTS:
Time Frame: From first dose of denosumab in Study 20110113 to end of study. Median (minimum, maximum) time on study was 13.93 (0.0, 74.7) months.
Description: Other Adverse Events summarizes the non-serious occurrences of adverse events that exceed the indicated frequency threshold.
Arm/Group | Denosumab
All-Cause Mortality (participants affected / at risk) | 18/128
Serious Adverse Events (participants affected / at risk) | 45/128
Other Adverse Events (participants affected / at risk) | 66/128
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Denosumab (N=128)
Anaemia (Blood and lymphatic system disorders) | 3
Febrile neutropenia (Blood and lymphatic system disorders) | 2
Arrhythmia (Cardiac disorders) | 1
Cardiac arrest (Cardiac disorders) | 1
Cardiac failure (Cardiac disorders) | 1
Cardiopulmonary failure (Cardiac disorders) | 1
Abdominal pain (Gastrointestinal disorders) | 2
Ascites (Gastrointestinal disorders) | 2
Intestinal obstruction (Gastrointestinal disorders) | 2
Melaena (Gastrointestinal disorders) | 1
Nausea (Gastrointestinal disorders) | 1
Vomiting (Gastrointestinal disorders) | 2
Asthenia (General disorders) | 1
Disease progression (General disorders) | 2
General physical health deterioration (General disorders) | 2
Cholecystitis acute (Hepatobiliary disorders) | 1
Jaundice (Hepatobiliary disorders) | 1
Abscess jaw (Infections and infestations) | 1
Cellulitis (Infections and infestations) | 1
Myelitis (Infections and infestations) | 1
Osteomyelitis (Infections and infestations) | 3
Pneumonia (Infections and infestations) | 4
Pulpitis dental (Infections and infestations) | 1
Septic shock (Infections and infestations) | 1
Upper respiratory tract infection (Infections and infestations) | 1
Fall (Injury, poisoning and procedural complications) | 1
Femur fracture (Injury, poisoning and procedural complications) | 1
Cachexia (Metabolism and nutrition disorders) | 2
Hypoglycaemia (Metabolism and nutrition disorders) | 1
Muscle spasms (Musculoskeletal and connective tissue disorders) | 1
Muscular weakness (Musculoskeletal and connective tissue disorders) | 1
Osteonecrosis of jaw (Musculoskeletal and connective tissue disorders) | 7
Breast cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2
Cardiac myxoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Metastases to liver (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Neoplasm malignant (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Prostate cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2
Hemiparesis (Nervous system disorders) | 1
Paraplegia (Nervous system disorders) | 1
Radiculopathy (Nervous system disorders) | 1
Vertebrobasilar insufficiency (Nervous system disorders) | 1
Acute kidney injury (Renal and urinary disorders) | 1
Acute pulmonary oedema (Respiratory, thoracic and mediastinal disorders) | 1
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 1
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 3
Pleurisy (Respiratory, thoracic and mediastinal disorders) | 1
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 2
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Denosumab (N=128)
Anaemia (Blood and lymphatic system disorders) | 8
Abdominal pain (Gastrointestinal disorders) | 9
Diarrhoea (Gastrointestinal disorders) | 11
Nausea (Gastrointestinal disorders) | 15
Toothache (Gastrointestinal disorders) | 9
Vomiting (Gastrointestinal disorders) | 11
Asthenia (General disorders) | 15
Fatigue (General disorders) | 12
Decreased appetite (Metabolism and nutrition disorders) | 14
Arthralgia (Musculoskeletal and connective tissue disorders) | 15
Back pain (Musculoskeletal and connective tissue disorders) | 16
Osteonecrosis of jaw (Musculoskeletal and connective tissue disorders) | 8
Pain in extremity (Musculoskeletal and connective tissue disorders) | 13
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 7

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The Clinical Trial Agreement generally does not restrict an investigator's discussion of trial results after completion. The Agreement permits Amgen a limited period of time to review material discussing trial results (typically up to 45 days and possible extension). Amgen may remove confidential information, but authors have final control and approval of publication content. For multicenter studies, the investigator agrees not to publish any results before the first multi-center publication.

DOCUMENTS (2):
  • Study Protocol (2013-02-22): https://cdn.clinicaltrials.gov/large-docs/17/NCT01419717/Prot_000.pdf
  • Statistical Analysis Plan (2018-08-27): https://cdn.clinicaltrials.gov/large-docs/17/NCT01419717/SAP_001.pdf